CLINICAL TRIAL: NCT02113761
Title: Non Invasive Mapping Before Ablation for Atrial Fibrillation: the Afacart Study.
Brief Title: Non Invasive Mapping Before Ablation for Atrial Fibrillation.
Acronym: AFACART
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Collaborators: Centre Hospitalier Universitaire Brugmann (Other)
Responsible Party: Principal Investigator, Pr Sébastien Knecht, PMD PhD, Brugmann University Hospital
Other Study IDs: BE77201318160
Record Dates: First submitted 2014-03-19; First posted 2014-04-15 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
RATIONALE / CONTEXT The ECG records the electrical activity propagating along cardiac cells (from the atria to the ventricles). The standard 12 ECG leads placed on the chest measure the global activation of the heart and do not have the ability to detect small-scale disturbances or to pinpoint ectopic activity. By the 1960s, multiple electrodes were placed around the chest to try to understand the complexity of the distribution of electrical activity in relation to the single cardiothoracic geometry of each individual. The safety of this method is similar to the ECG but its superiority has been demonstrated by the detection of anomalies imperceptible to the standard ECG. The accuracy of the technique in localizing rhythm disturbances is on the order of 5 mm.

OBJECTIVES Main objective: To evaluate the utility of noninvasive mapping during persistent AF electrophysiology procedure

Secondary objectives:

1. Compare the effectiveness of noninvasive mapping compared to conventional standard of care methods for AF mapping and ablation procedure.
2. Evaluate the absence of recurrence of persistent AF after a follow up of 12 months after the procedure during a scheduled hospitalization.

DIAGRAM OF RESEARCH European Diagnostic Study, feasibility, non-randomized, multi center

RESEARCH PROCEDURES A trained clinical specialist places 252 dry gelled ECG electrodes on the patient's torso. The 252 ECG electrode array is hooked up to the CardioInsight system and body surface ECG recordings are made during the patient's arrhythmia. The patient is then sent to the radiology department for a CT scan (no contrast) to image both the heart and electrodes on the patient's torso. A trained clinical specialist from CardioInsight then segments the CT DICOM images from the CT scan to obtain epicardial anatomy and establish heart-torso geometry.

The electrograms are processed by the system to produce movies of fibrillatory activity (both focal activity, and rotor activity).

PROCEDURAL ENDPOINTS Primary endpoint: Acute AF termination to atrial tachycardia or sinus rhythm

Secondary outcome criteria:

* Reduction in RF time compared to standard of care (historical control - comparable patient population)
* Reduction in procedure time compared to standard of care (historical control - comparable patient population)
* Freedom from persistent AF at the end of the 12 months F/U period STUDY SIZE

The sample size was estimated at 100 patients, with up to 20 patients per center STUDY CENTERS 8 Centers :

* Brugmann - Brussels (Belgium)
* Clinique Pasteur - Toulouse (France)
* Medizinische Klinik und Poliklinik - Mainz (Germany)
* University ed Herzzentrum Freiburg Bad Kozingen (Germany)
* Deutsches Herzzentrum München, Munich (Germany)
* Kerkhoff Klinik, Bad Nauheim, (Germany)
* Sint-Jan Sint-Franciscus Xaverius, Brugge (Belgium)
* Clinique Ambroise Paré, Paris, France

EXPECTED OUTCOME In patients referred for ablation of persistent AF, ECG mapping data will be correlated to the invasive procedure. It is expected that procedure time will be statistically shorter and total RF energy delivery is expected to be smaller than that of standard of care for AF treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female Adults (≥18 years old)
* Minors (15-18 years) of both sexes subject to parental consent or legal representative
* Persistent AF ablation refractory to drugs
* Persistent AF (as defined by consensus statement) for ≤ 12 month duration
* Consent signed by the patient after reading the information leaflet

Exclusion Criteria:

* Any previous left atrial (LA) ablation
* Any previous LA or RA surgery
* Current intra-cardiac thrombus
* Presence of any pulmonary vein stents
* Presence of any pre-existing pulmonary vein stenosis
* Anteroposterior LA diameter > 5.5 cm by TTE or CT
* Presence of any cardiac valve prosthesis
* Clinically significant mitral valve regurgitation or stenosis
* Myocardial infarction, PCI / PTCA or coronary artery stenting within the last 3 months
* Unstable angina
* Any cardiac surgery within the last 3 months
* NYHA class III or IV congestive heart failure
* Uncontrolled hyperthyroidism
* Any cerebral ischemic event (strokes or TIAs) which occurred during the 6 months interval preceding the consent Date.
* Life expectancy less than one (1) year
* Current or anticipated participation in any other clinical trial of a drug, device or biologic should be done only after prior consultation and approval of the investigator(s)
* Unwilling or unable to comply fully with study procedures and follow-up

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with persistent atrial fibrillation as described by the Consensus Statement and with an indication for atrial fibrillation catheter ablation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
radiofrequency duration | 1 day (At the end of the procedure)
  Radiofrequency duration necessary to terminate atrial fibrillation and total radiofrequency duration
Atrial fibrillation termination | At the time of the procedure of catheter ablation
  Amount of patients with AF termination into sinus rhythm or atrial tachycardia during AF ablation.

SECONDARY OUTCOMES:
Atrial fibrillation recurrence | One year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brugmann, Brussels, Belgium